CLINICAL TRIAL: NCT00684827
Title: A Cumulative Dose Tolerability Study of Levalbuterol HFA and Racemic Albuterol HFA in Subjects Twelve Years of Age and Older With Asthma
Brief Title: A Safety and Tolerability Study of Levalbuterol HFA Metered Dose Inhaler in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 051-310
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Asthma; Racemic albuterol
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects will receive both treatments: (a) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses); followed by (b) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses).
  The first treatment will be administered, followed by a 7 ±2 days washout period, after which the second of the two treatments will be administered. Cumulative dosing will occur according to the following schedule: 1 puff at 0 and 30 minutes, 2 puffs at 60 minutes, 4 puffs at 90 minutes and 8 puffs at 120 minutes. An AeroChamber Plus spacer will be utilized for each dose
  Interventions: Drug: Levalbuterol HFA MDI followed by Racemic albuterol HFA MDI
- B (Active Comparator): Subjects will receive both treatments: (a) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses) followed by (b) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses) The first treatment will be administered, followed by a 7 ±2 days washout period, after which the second of the two treatments will be administered. Cumulative dosing will occur according to the following schedule: 1 puff at 0 and 30 minutes, 2 puffs at 60 minutes, 4 puffs at 90 minutes and 8 puffs at 120 minutes. An AeroChamber Plus spacer will be utilized for each dose.
  Interventions: Drug: Racemic Albuterol followed by levalbuterol HFA MDI

INTERVENTIONS:
Drug: Levalbuterol HFA MDI followed by Racemic albuterol HFA MDI — 1. Subjects will receive both treatments: (a) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses); followed by (b) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses)
  2. Arm #A
  3. Xopenex HFA MDI, Pirbuterol HFA MDI
  Arms: A
Drug: Racemic Albuterol followed by levalbuterol HFA MDI — 1. Subjects will receive both treatments: (a) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses) followed by (b) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses)
  2. Arm #B
  3. Pirbuterol HFA MDI, Xopenex HFA MDI
  Arms: B

SUMMARY:
The purpose of this study is to compare the safety and tolerability of levalbuterol HFA metered dose inhaler (MDI) versus racemic albuterol HFA MDI.

DETAILED DESCRIPTION:
A randomized, modified-blind active-controlled multicenter, two-way crossover study of levalbuterol compared to racemic albuterol (using a spacer) in subjects 12 years of age and older with asthma. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, must be at least 12 years of age at the time of consent.
* Female subjects 12-60 years of age inclusive must have a negative serum pregnancy test at study start.
* Women of child bearing potential must be using an acceptable method of birth control throughout the study.
* Subject must have a documented diagnosis of asthma for a minimum of 6 months prior to study start.
* Subject must be in good health with the exception of their reversible airways disease and not suffering from any chronic condition that might affect their respiratory function.
* Subject must have a chest X-ray or had one within 12 months prior to randomization.
* Subject must be able to complete the diary cards and medical event calendars reliably on a daily basis, understand dosing instructions and be able to demonstrate good MDI administration technique. Any minor subject who is not able to do this must have a parent/legal guardian who can assist them during the study with these activities.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Subject who has participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another clinical trial.
* Subject whose schedule prevents him or her from starting study visits before 9 AM.
* Subject who has travel commitments during the study that would interfere with trial measurements or compliance or both.
* Subject who has a history of hospitalization for asthma within 4 weeks prior to study start, or who is scheduled for in-patient hospitalization, including elective surgery during the course of the trial
* Subject with a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations.
* Subject using any prescription drug with which albuterol sulfate administration is contraindicated.
* Subject with currently diagnosed life-threatening asthma defined as a history of asthma episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures within 12 months prior to study start.
* Subject with a history of cancer (exception: basal cell carcinoma in remission).
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders.
* Subject with a history of substance abuse or drug abuse within 12 months preceding study start.
* Subject with greater than 10 pack year history of cigarette smoking or use of any tobacco products within 6 months of study start.
* Subject with a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis.
* Subject who has suffered from a clinically significant upper or lower respiratory tract infection in the 3 weeks prior to study start.
* Subject with unstable asthma; or who have had a change in asthma therapy; or a visit to the Emergency Department or hospital for worsening asthma within 4 weeks.
* Subject who is a staff member or relative of a staff member.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-10; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Increases from visit pre-dose to each post-dose dose measurement in heart rate, blood pressure (systolic and diastolic), potassium and glucose | Days 0, 7, 10

SECONDARY OUTCOMES:
Percent change in FEV1 (from visit pre-dose to each post dose measure) | Days 0, 7, 10
Percent change in FVC (from visit pre-dose to each post dose measure); | Days 0, 7, 10
Percent change in FEF25-75% (from visit pre-dose to each post dose measure); | Days 0, 7, 10
Number of cumulative actuations received | Days 0, 7, 10

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Encinitas, California
  - Los Angeles, California
  - North Dartmouth, Massachusetts
  - St Louis, Missouri